CLINICAL TRIAL: NCT04571320
Title: A Peer-Delivered High School Preparatory Intervention for Students With ADHD
Acronym: Summer STRIPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Margaret Sibley, Associate Professor of Psychiatry & Behavioral Health, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH122225 (NIH); R34MH122225 (NIH)
Record Dates: First submitted 2020-08-31; First posted 2020-10-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: ADHD
Keywords: ADHD; School-based; Peer-delivered; Adolescence
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Teachers and outcomes assessors will be masked to group; however, it will not be possible to mask parents and adolescents to group because they will be actively receiving a behavioral intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Summer STRIPES (Experimental): Up to two weeks of daily high school orientation (four hours per day) immediately prior to the start of ninth grade, staffed by peer interventionists (2:1 ratio + extra interventionist in case of absences) and a school staff member. Two sessions of summer parent training. During the school year, ninth grade students will continue to meet weekly with their peer interventionists in a group setting under the supervision of the school staff sponsor. School year follow-up component of summer STRIPES will occur for 16 weeks and will include weekly 30 minute meetings between peer and target students. Parent components during the school year will include optional monthly group problem solving sessions with the school staff sponsor and school mental health liaison and a weekly phone call (up to five minutes) from the school staff sponsor to discuss home contingency management.
  Interventions: Behavioral: Summer STRIPES
- Enhanced School Services as Usual (Active Comparator): Students who are assigned to the SSU plus group will be referred to their identified school counselor for referral to services available in the school setting. The counselor will be provided with a report from the student's intake assessment that summarizes the student's symptoms and presenting problems. The student will also receive new school supplies at the beginning of ninth grade. In our past trials, SSU plus students typically received subject-specific tutoring or after-school homework help. We will systematically track services received by students in the SSU plus condition.
  Interventions: Other: Enhanced School Services as Usual

INTERVENTIONS:
Behavioral: Summer STRIPES — See arm description.
  Arms: Summer STRIPES
Other: Enhanced School Services as Usual — see arm description.
  Other Names: SSU plus
  Arms: Enhanced School Services as Usual

SUMMARY:
This study will test whether a peer-delivered intervention for high school students with ADHD outperforms enhanced school services as usual. Ninth grade students with ADHD (N=72) will be randomly assigned to the intervention (summer STRIPES) or the enhanced school services control group (SSU plus). Students will be assessed in the spring of 8th grade, fall of ninth grade, and spring of ninth grade. Primary outcomes will be GPA, Class Attendance, Disciplinary Incidents, and ADHD symptoms (parent and teacher report).

DETAILED DESCRIPTION:
The proposed study will adapt and test a low resource school-based intervention to prepare students with ADHD for the transition to high school-a point of vulnerability for youth with ADHD. The resulting intervention will be delivered as a peer-delivered orientation to high school (1-2 weeks for 4 hours a day) with weekly peer-delivered support during the first 16 weeks of the ninth grade year. Intervention development will involve scaling down an intensive Summer Treatment Program for adolescents with ADHD, using its core components (i.e., daily skills training and repetition, parent coaching in contingency management, engaging recreational activities) to bolster a promising peer-delivered school-based intervention for ninth graders with ADHD. The resulting intervention (summer STRIPES) will target three mechanisms that are critical markers of high school success: (a) intrinsic motivation, (b) extrinsic motivation, and (c) executive functions (EFs). Y01, will use a stakeholder informed process to iteratively adapt the intervention with input from two partnering high schools (i.e., administrators, counselors, teachers, parents, students) and content experts (Sibley, Langberg, Sasser, Aaronson). Two manuals that are individualized for each school will emerge. A total of 72 rising ninth grade students with ADHD will be recruited in Y02 and Y03 (36 per year; 18 per school) from two high schools randomly assigned (within school) to receive summer STRIPES or enhanced school services as usual (SSU plus). A school staff summer STRIPES sponsor at each school will oversee training and supervision peer interventionists with support from investigators. Peer interventionists will receive a three-day training and weekly supervision. Study assessments will occur at baseline and three follow-up points throughout the ninth grade year. To test the intervention's preliminary effectiveness, the study will examine treatment effects on GPA, class attendance, and disciplinary incidents. Preliminary effectiveness will also be measured through indices of engagement (parent, adolescent, peer attendance, ratings of satisfaction, perceived utility, and therapeutic alliance) and school fit (treatment fidelity, peer attitudes toward treatment). To detect whether therapeutic mechanisms (intrinsic motivation, extrinsic motivation, EFs) are engaged by summer STRIPES, the investigators will test for group differences on multi-method indices of these mechanisms, as well as the extent to which hypothesized mechanisms affect meaningful change on study outcomes. This project represents the first attempt to utilize a peer-delivered model for ADHD intervention in a high school orientation context. If summer STRIPES participants show meaningful improvements in functioning and engagement and school fit are strong, an R01 will be planned to fully evaluate the effectiveness of this approach. To inform this future trial, attention will be given to developing an optimal measurement battery, treatment delivery model, and recruitment strategy for rising ninth graders.

ELIGIBILITY:
Inclusion Criteria:

* Meet Symptom and Impairment Criteria for DSM-5 ADHD
* Attending ninth grade at a participating school

Exclusion Criteria:

* Placement in special education classes
* IQ < 70

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Grade Point Average | Change from Baseline to End of 9th grade, an average of 1 year
  Quarterly Student Grade Point Average from Report Cards
Class Attendance | Change from Baseline to End of 9th grade, an average of 1 year
  Number of Class Absences per Academic Quarter
Attention Deficit Hyperactivity Disorder Symptom Severity | Change from Baseline to End of 9th grade, an average of 1 year
  Parent and Teacher Rated ADHD Symptoms on DSM-5 ADHD Checklist, 0=minimum, 3=maximum, Higher score means worse outcome

OTHER OUTCOMES:
Target Mechanism: Extrinsic Motivation (measure 1) | Change from Baseline to End of 9th grade, an average of 1 year
  Expectancy Value Theory of Motivation Measure (Student Report); Importance Subscale
  1=minimum, 5=maximum, higher scores mean better outcome
Target Mechanism: Extrinsic Motivation (measure 2) | Change from Baseline to End of 9th grade, an average of 1 year
  Hungry Donkey Task (IOWA Gambling Task) --Risky Decision Making
Target Mechanism: Extrinsic Motivation (measure 3) | Change from Baseline to End of 9th grade, an average of 1 year
  Delay Discounting measured on Choice Delay task (total amount of money earned)
Target Mechanism: Extrinsic Motivation (measure 4) | Change from Baseline to End of 9th grade, an average of 1 year
  The Change Ruler self-report, 1=minimum value 10=maximum value, higher scores mean better outcome
Target Mechanism: Intrinsic Motivation (measure 1) | Change from Baseline to End of 9th grade, an average of 1 year
  Expectancy-Value Theory of Motivation Measure-Student Version, Interest subscale, 1=minimum, 5=maximum, higher scores mean better outcome
Target Mechanism: Intrinsic Motivation (measure 2) | Change from Baseline to End of 9th grade, an average of 1 year
  Delay Aversion; Quick Delay Questionnaire (self-report), 1=minimum value 5=maximum value, higher scores better outcomes, items 5-10 reverse coded
Target Mechanism: Intrinsic Motivation (measure 3) | Change from Baseline to End of 9th grade, an average of 1 year
  Change Ruler Scale self-report, 1=minimum value 10=maximum value, higher scores mean better outcome
Target Mechanism: Intrinsic Motivation (measure 4) | Change from Baseline to End of 9th grade, an average of 1 year
  Basic Psychological Needs Scale self-report, 1=minimum value 6=maximum value, higher scores mean better outcome
Target Mechanism: Executive Functions (measure 1) | Change from Baseline to End of 9th grade, an average of 1 year
  parent report: goal setting and planning section of the Self-Regulated Learning Interview Schedule
Target Mechanism: Executive Functions (measure 2) | Change from Baseline to End of 9th grade, an average of 1 year
  Behavior Rating Index of Executive Function (BRIEF-2) parent report
Target Mechanism: Executive Functions (measure 3) | Change from Baseline to End of 9th grade, an average of 1 year
  National Institute of Health (NIH) Toolbox List Sorting Working Memory Test
Target Mechanism: Executive Functions (measure 4) | Change from Baseline to End of 9th grade, an average of 1 year
  go/no-go task (number of commission errors on no-go trials)
Target Mechanism: Executive Functions (measure 5) | Change from Baseline to End of 9th grade, an average of 1 year
  NIH Toolbox Dimensional Change Card Sort Test
Target Mechanism: Executive Functions (measure 6) | Change from Baseline to End of 9th grade, an average of 1 year
  observations of planner use (or a device if preferred)
Target Mechanism: Executive Functions (measure 7) | Change from Baseline to End of 9th grade, an average of 1 year
  bookbag organization. Percentage of classes with recorded homework (or indication of no homework) will be calculated for the last five school days
Target Mechanism: Executive Functions (measure 8) | Change from Baseline to End of 9th grade, an average of 1 year
  note-taking skills analogue paradigm
Target Mechanism: Executive Functions (measure 9) | Change from Baseline to End of 9th grade, an average of 1 year
  Adolescent Academic Problems Checklist
Engagement and Fit Measures: Fidelity Checklists | During Intervention Delivery, an average of 1 year
  % of fidelity items marked yes for treatment and supervision sessions
Engagement and Fit Measures: Intervention Attendance | During Intervention Delivery, an average of 1 year
  % of intervention sessions attended by student and peers and parents
Engagement and Fit Measures: Parent Academic Involvement | Change from Baseline to End of 9th grade, an average of 1 year
  Parent Academic Management Scale (PAMS) completed by parent, 0=minimum value 5=maximum value, higher scores mean better outcome
Engagement and Fit Measures: Intervention Credibility | Immediately post-treatment
  Client Credibility Questionnaire completed by student,and peer interventionist, 0=minimum value 2=maximum value, Higher scores mean a better outcome
Engagement and Fit Measures: Intervention Credibility | Immediately post-treatment
  Client Credibility Questionnaire completed by parent, 0=minimum value 8=maximum value, Higher scores mean a better outcome
Engagement and Fit Measures: Satisfaction | Immediately post-treatment
  STRIPES Satisfaction Questionnaire completed by student, peer interventionist, and parent, 1=minimum value 5=maximum value, higher scores mean better outcome
Engagement and Fit Measures: Therapy-Bond and Engagement Scales | Immediately post-treatment
  Therapy Bond and Engagement Scale completed by student and peers, 1=minimum 4=maximum, higher scores means better outcome
Follow-up Focus Groups and Surveys | Immediately post-treatment
  Qualitative data collected from parents
Follow-up Focus Groups and Surveys | Immediately post-treatment
  Qualitative data collected from peers
Follow-up Focus Groups and Surveys | Immediately post-treatment
  Qualitative data collected from students
Time Varying Covariate: Medication Use | Change from Baseline to End of 9th grade, an average of 1 year
  Medication Use Interview

CONTACTS AND LOCATIONS:
Overall Officials: Margarret Sibley, Ph.D., Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Zulauf-McCurdy CA, Coxe SJ, Lyon AR, Aaronson B, Ortiz M, Sibley MH. Study protocol of a randomised trial of Summer STRIPES: a peer-delivered high school preparatory intervention for students with ADHD. BMJ Open. 2021 Aug 3;11(8):e045443. doi: 10.1136/bmjopen-2020-045443. PMID 34344674